CLINICAL TRIAL: NCT04035005
Title: A Phase IIIb Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Ocrelizumab in Adults With Primary Progressive Multiple Sclerosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Ocrelizumab in Adults With Primary Progressive Multiple Sclerosis
Acronym: O'HAND
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA40404; 2018-001511-73 (EudraCT Number); 2023-505980-36-00 (EU CTIS Number)
Record Dates: First submitted 2019-07-17; First posted 2019-07-29 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab (Experimental): Participants will receive ocrelizumab by intravenous (IV) infusion every 24 weeks.
  Interventions: Drug: Ocrelizumab
- Placebo (Placebo Comparator): Participants will receive placebo matched to ocrelizumab by IV infusion every 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocrelizumab — The first dose of ocrelizumab will be administered as two 300 milligrams (mg), IV infusions given 14 days apart. For the subsequent doses, ocrelizumab will be administered as a single 600 mg infusion every 24 weeks. A minimum interval of 20 or 22 weeks, depending on if the previous dose was administered in one or two infusion, should be maintained between each infusion.
  Other Names: Ocrevus
  Arms: Ocrelizumab
Drug: Placebo — The first dose of placebo will be administered as two IV infusions given 14 days apart. For the subsequent doses, placebo will be administered as a single infusion every 24 weeks, with a minimum interval of 20 or 22 weeks, depending on if the previous dose was administered in one or two infusions, maintained between each infusion.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ocrelizumab (Ocrevus®) compared with placebo in participants with primary progressive multiple sclerosis (PPMS), including participants later in their disease course. This study will consist of the following phases: screening, double-blind treatment, an optional post-double-progression ocrelizumab (PDP OCR) treatment, follow-up 1 (FU1), an optional open-label extension (OLE), and follow-up 2 (FU2).

DETAILED DESCRIPTION:
The screening phase will last up to 24 weeks. In the double-blind treatment phase, participants will undergo at least 144 weeks of study treatment. Study drug (ocrelizumab or placebo) will be administered every 24 weeks. All participants who discontinue prematurely from the double-blind treatment phase will enter the FU1 phase, including participants receiving other immunomodulatory or immunosuppressive treatment(s) for MS, commercial ocrelizumab, or no treatment. The FU1 phase will run in parallel with the double-blind treatment phase for 144 weeks or until the primary analysis is performed, whichever occurs first. An optional OLE phase is planned for eligible participants who either have either completed 144 weeks of the double-blind treatment phase or are ongoing in the double-blind treatment phase at the time of the primary analysis and, in the opinion of the investigator, could benefit from ocrelizumab treatment. The following participants will move into the FU2 phase: participants who are ongoing in the FU1 at 144 weeks from randomization or at the time of the primary analysis; participants who have either completed 144 weeks of the double-blind treatment phase or are ongoing in the double-blind treatment phase at the time of the primary analysis and will not enter the OLE phase; participants who have completed or withdrawn from the OLE phase or from PDP OCR treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* EDSS score at screening and baseline >= 3.0 to 8.0, inclusive
* Disease duration from the onset of MS symptoms relative to randomization date:

Less than 20 years in participants with an EDSS score at screening 7.0 - 8.0 Less than 15 years in participants with an EDSS at screening 5.5 - 6.5 Less than 10 years in participants with an EDSS at screening <= 5.0

* Documented history or presence at screening of at least one of the following laboratory findings in a cerebrospinal fluid specimen: Elevated immunoglobulin G (IgG) index or one or more IgG oligoclonal bands detected by isoelectric focusing
* Screening and baseline 9-HPT completed in > 25 seconds (average of the two hands)
* Neurological stability for ≥ 30 days prior to baseline
* Ability to complete the 9-HPT within 240 seconds with each hand at screening and baseline
* Neurological stability for >/= 30 days prior to baseline
* Participants previously treated with immunosuppressants, immunomodulators, or other immunomodulatory therapies must undergo an appropriate washout period according to the local label of the immunosuppressant/immunomodulatory drug used
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraceptive methods during the treatment period and for 6 or 12 months after the final dose of ocrelizumab. Adherence to local requirements, if more stringent, is required.
* For female participants without reproductive potential: Women may be enrolled if surgically sterile (i.e hysterectomy, complete bilateral oophorectomy) or post-menopausal unless the participant is receiving a hormonal therapy for her menopause or if surgically sterile

Exclusion Criteria:

* History of relapsing-remitting or secondary progressive MS at screening
* Confirmed serious opportunistic infection including: active bacterial, viral, fungal, mycobacterial infection or other infection, including tuberculosis or atypical mycobacterial disease
* Participants who have or have had confirmed or a high degree of suspicion of progressive multifocal leukoencephalopathy (PML)
* Known active malignancy or are being actively monitored for recurrence of malignancy
* Immunocompromised state
* Receipt of a live-attenuated vaccine within 6 weeks prior to randomization
* Inability to complete an MRI or contraindication to Gd administration.
* Participants requiring symptomatic treatment of MS and/or physiotherapy who are not on a stable regimen. Participants must not initiate symptomatic treatment of MS or physiotherapy within 4 weeks of randomization.
* Contraindications to mandatory premedications for infusion-related reactions, including:

uncontrolled psychosis for corticosteroids and closed-angle glaucoma for antihistamines

* Known presence of other neurologic disorders
* Pregnant or breastfeeding, or intending to become pregnant during the study and for 6 or 12 months after last infusion of the study drug
* Lack of peripheral venous access
* Significant, uncontrolled disease, such as cardiovascular, pulmonary, renal, hepatic, endocrine or gastrointestinal, or any other significant disease that may preclude participant from participating in the study
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History of alcohol or other drug abuse
* History of primary or secondary immunodeficiency
* Treatment with any investigational agent within 24 weeks prior to screening (Visit 1) or 5 half-lives of the investigational drug (whichever is longer), or treatment with any experimental procedure for MS
* Previous treatment with B-cell targeting therapies
* Any previous treatment with bone marrow transplantation and hematopoietic stem cell transplantation
* Any previous history of transplantation or anti-rejection therapy
* Treatment with IV Ig or plasmapheresis within 12 weeks prior to randomization
* Systemic corticosteroid therapy within 4 weeks prior to screening
* Positive serum human chorionic gonadotropin (hCG) measured at screening or positive urine β-hCG at baseline
* Positive screening tests for hepatitis B
* Any additional exclusionary criterion as per ocrelizumab (Ocrevus®) local label, if more stringent than the above
* Lack of MRI activity at screening/baseline if more than 650 participants without MRI activity have already been enrolled, as defined by T1 Gd+ lesion(s) and/or new and/or enlarged T2 lesion(s) in the screening, to ensure that at least 350 participants with MRI activity will be randomized

Eligibility Criteria for OLE Phase:

* Completed the 144 weeks of double-blind treatment phase of the trial or are ongoing in the double blind treatment phase at the time of the primary analysis, and who, in the opinion of the investigator, may benefit from treatment with Ocrelizumab. Participants who withdrew from study treatment and received another DMT or commercial ocrelizumab will not be allowed to enter in the OLE phase.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use adequate contraceptive methods during the treatment period and for 6 or 12 months after the final dose of ocrelizumab. Adherence to local requirements, if more stringent, is required.
* For female participants without reproductive potential: Women may be enrolled if surgically sterile (i.e. hysterectomy, complete bilateral oophorectomy) or post-menopausal unless the participant is receiving a hormonal therapy for her menopause or if surgically sterile

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2028-01-19 (Estimated)

PRIMARY OUTCOMES:
Time to Onset of Composite 12-week Confirmed Disability Progression (CDP) | Baseline up to approximately 144 weeks

SECONDARY OUTCOMES:
Time to 12-week CDP in 9-Hole Peg Test (9-HPT) | Baseline up to approximately 144 weeks
  The 9-HPT is a quantitative measure of upper extremity (arm and hand) function (Goodkin et al. 1988; Fischer et al. 1999b).
Time to 12-week CDP in EDSS | Baseline up to approximately 144 weeks
  Disability progression was measured by EDSS and is defined as an increase of ≥1 point from baseline EDSS score in participants with a baseline EDSS score ≤ 5.5 or an increase of ≥ 0.5 point in participants with a baseline EDSS score of < 5.5 that is confirmed for at least 12 weeks. The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
Time to 24-week CDP in 9-HPT | Baseline up to approximately 144 weeks
  The 9-HPT is a quantitative measure of upper extremity (arm and hand) function (Goodkin et al. 1988; Fischer et al. 1999b).
Time to 24-week CDP in EDSS | Baseline up to approximately 144 weeks
  Disability progression was measured by EDSS and is defined as an increase of ≥1 point from baseline EDSS score in participants with a baseline EDSS score ≤ 5.5 or an increase of ≥ 0.5 point in participants with a baseline EDSS score of < 5.5 that is confirmed for at least 12 weeks. The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
Annual Rate of Percent Change From Baseline in Total Volume of T2 Lesions on Magnetic Resonance Imaging (MRI) Scans | Baseline up to approximately 8.5 years
Annual Rate of Percent Change From 24 Week in Total Brain Volume on MRI Scans | Week 24 up to approximately 8.5 years
Percentage of Participants with Adverse Events (AEs) | Up to approximately 8.5 years
Percentage of Participants With Serious Adverse Events (SAEs) | Up to approximately 8.5 years
Percentage of Participants With AEs Leading to Study Treatment Withdrawal | Up to approximately 8.5 years
Number of Participants With Anti-Drug Antibodies (ADAs) to Ocrelizumab | Up to approximately 8.5 years
Plasma Concentration of Ocrelizumab | Baseline, Weeks 2, 12, 24, 48, 60, 72, and every 12 weeks till the end of the double-blind period and Weeks 0 and 48 of the OLE period
Evaluation of Ocrelizumab Pharmacodynamics, as Measured by B-Cell Levels in Blood | Baseline, Weeks 2, 24, 48, 72 and every 12 weeks till the end of the double-blind period and Weeks 0, 22, 46, 70 and 96 of the OLE period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (159):
- United States (11):
  - Multiple Sclerosis Center of California, Laguna Hills, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MS and Neuromuscular Center of Excellence, Clearwater, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Vero Neurology, Vero Beach, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Michigan Neurology Associates P.C., Clinton Township, Michigan
  - The Boster Center for MS, Columbus, Ohio
  - Columbus Neuroscience, Westerville, Ohio
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Maxine Mesinger MS Clinic/Baylor College of Medicine, Houston, Texas
- Australia (3):
  - Brain and Mind Research Institute, Camperdown, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (3):
  - UZ Antwerpen, Edegem, Antwerpen
  - Cliniques Universitaires St-Luc, Brussels
  - MS & Neurologisch Revalidatie Centrum, Overpelt
- Bulgaria (3):
  - Military Medical Academy HBAT, Pleven
  - Multiprofile Hospital For Active Treatment Avis Medica, Pleven
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry Sv. Naum EAD, Sofia
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Dalhousie Multiple Sclerosis Research Unit, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
  - Recherche Sepmus Inc., Greenfield Park, Quebec
- Colombia (2):
  - Instituto Neurologico de Colombia INDEC, Medellín, Antioquia
  - Clinica Colsanitas S.A. sede Clinica Universitaria Colombia, Bogotá
- Croatia (4):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Sestre Milosrdnice, Zagreb
  - University Hospital Center Zagreb, Zagreb
- France (6):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire de Clermont Ferrand, Clermont-Ferrand
  - CHRU Nancy, Nancy
  - Hopital Guillaume Et Rene Laennec, Nantes
  - CHU de Nimes - Hopital Universitaire Caremeau, Nîmes
  - Hopital Civil, Strasbourg
- Georgia (3):
  - Pineo Medical Ecosystem LTD, Tbilisi
  - The First University Clinic of Tbilisi State Medical University, Tbilisi
  - Khechinashvili University Hospital, Tbilisi
- Italy (8):
  - AOU dell Universita degli Studi della Campania Luigi Vanvitelli Piazza Luigi Miraglia 2, Napoli, Campania
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Azienda Ospedaliera Sant'andrea, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Fondazione Istituto G. Giglio di Cefalu, Cefalù, Sicily
- Lebanon (2):
  - Hotel Dieu de France, Achrafieh Beirut
  - Saint George University Medical Hospital, El Achrafiyé
- Mexico (5):
  - Grupo Medico Camino, Mexico City, Mexico CITY (federal District)
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Hospital Angeles Chihuahua, Chihuahua City
  - Unidad de Investigacion en Salud de Chihuahua, Mexico City
  - Clinical Research Institute, Tlalnepantla
- Morocco (2):
  - CHU Mohammed VI, Marrakesh
  - Centre Hospitalier Ibn Sina CHIS - Hopital des Specialites, Rabat
- New Zealand (2):
  - New Zealand Clinical Research - Christchurch, Christchurch
  - Dunedin Hospital, Dunedin
- Poland (20):
  - Neurocentrum Bydgoszcz sp z o.o, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Przychodnia EuroMediCare, Wroclaw, Lower Silesian Voivodeship
  - Rejdak Konrad Indywidualna Praktyka Lekarska dr hab. Konrad Rejdak, Lublin, Lublin Voivodeship
  - Centrum Medyczne Medyk, Rzeszów, Podkarpackie Voivodeship
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3, Rybnik, Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku Marii Sklodowskiej Curie 24a, Bia?ystok
  - Copernicus Podmiot Leczniczy Sp z o o, Gda?sk
  - Mazowieckie Centrum Badan Klinicznych, Grodzisk Mazowiecki
  - MA-LEK Clinical Sp. Z o.o., Katowice
  - Novo-Med Zielinski i wsp SpJ, Katowice
  - NEURO-MEDIC Sp. z o. o., Katowice
  - Specjalistyczna Praktyka Lekarska Dr n.med. Stanislaw Ochudlo, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Galen Clinic, Lublin
  - Wojewodzki Szpital Specjalistyczny, Olsztyn
  - Med-Polonia Sp. z o.o., Poznan
  - EUROMEDIS Sp z o o, Szczecin
  - Centrum Medyczne NeuroProtect Zablocinska 10, Warsaw
  - RESMEDICA Spolka z o.o., Kielce, Świętokrzyskie Voivodeship
- Portugal (5):
  - ULS de Loures-Odivelas, EPE - Hospital de Loures, Loures, Lisbon District
  - Hospital Garcia de Orta, Almada
  - Hospital de Braga, Braga
  - Hospital de Santo Antonio, Porto
  - Campus Neurologico Senior, Torres Vedras
- Romania (4):
  - Spitalul Judetean de Urgenta Deva, Deva, Hunedoara County
  - SC Clubul Sanatatii SRL, Campulung Muscel
  - Cai Ferate Clinical Hospital, Constanța
  - Targu Mures Clinical Emergency County Hospital, Târgu Mure?
- Russia (20):
  - Krasnoyarsk State Medical Academy, Krasnoyarsk, Krasnoyarsk Krai
  - City Clinical Hospital a n Buyanov V M, Moscow, Moscow Oblast
  - City Clinical Hospital #24, Moscow, Moscow Oblast
  - Moscow Regional Research Clinical Institute Na Mfvladimirskiy, Moscow, Moscow Oblast
  - Research Center of Neurology of RAMS, Moskva, Moscow Oblast
  - Neftyanik Medical and Sanitary Unit, Tumen, Moscow Oblast
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod, Niznij Novgorod
  - MEDIS Limited Liability Company, Nizhny Novgorod, Niznij Novgorod
  - SBHI of Nizhny Novgorod region City Clinical Hospital #3, Nizhny Novgorod, Niznij Novgorod
  - National Center of Socially Significant Diseases, Saint Petersburg, Sankt-Peterburg
  - City Hospital #40 of Kurortniy Administrative District, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital #4, Saransk, Saratov Oblast
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg, Sverdlovsk Oblast
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - Belyayev Clinical Hospital of the Kuzbass, Kemerovo
  - Kirov State Medical Academy, Kirov
  - FSBIH Siberian Regional Medical Centre of FMBA of Russia, Novosibirsk
  - Perm Regional Clinical Hospital of Znak Pocheta Medal, Perm
  - Siberian State Medical University of Roszdrav, Tomsk
- Serbia (7):
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia -PPDS, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Clinical Centre of Vojvodina, Nova Sad
  - General Hospital Uzice, Užice
- Spain (10):
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Complejo Asistencial Universitario de Salamanca ? H. Clinico, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Tunisia (4):
  - Hopital Razi, LA Mannouba
  - Fattouma Bourguiba University Hospital, Monastir
  - Hospital Habib Bourguiba, Sfax
  - Military Hospital of Tunis, Tunis
- Ukraine (21):
  - Treatment and diagnostic Center Neuro Global of LLC Neuro Global, Krykhivtsi, Ivano-Frankivsk Oblast
  - Communal noncommercial enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv, Kharkiv Governorate
  - Municipal Non-profit Enterprise Kherson City Clinical Hospital named after Ye.Ye. Karabelesh, Kherson, Kherson Governorate
  - Treatment and Diagnostic Center of LLC MRT Elit, Kropyvnytskyi, KIEV Governorate
  - Medical Centre of PE First Private Clinic, Kyiv, KIEV Governorate
  - Kyiv City Clinical Hospital #4, Kyiv, KIEV Governorate
  - Communal Non-Commercial Enterprise Clinical Hospital #15 of the Podilskyi District ofthe Kyiv City, Kyiv, KIEV Governorate
  - Municipal NPE Regional Clinical Center of Neurosurgery and Neurology of Transcarpathian RC, Uzhhorod, KIEV Governorate
  - Medical Center Artes Medicum LLC, Kyiv, Kyiv Oblast
  - Communal noncommercial enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Lviv, Lviv Oblast
  - Medical Center Salutem, Vinnytsia, Podolia Governorate
  - LLC Medical Center Health Clinic, Vinnytsia, Volhynian Governorate
  - LLC Medical Center Unimed, Zaporizhzhia, Zaporizhzhia Oblast
  - University hospital of Dnipro State Medical University, Dnipro
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Medical Center of LLC Medical Center Dopomoga Plus, Kyiv
  - Private Enterprise Clinic Medicom, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - LLC Medical Center INET 09, Zaporizhzhia
  - Municipal Non-profit Enterprise Zaporizhzhya Regional Hospital Zaporizhzhya Regional Council, Zaporizhzhia
- United Kingdom (10):
  - University Hospital of Wales, Cardiff
  - Queen Elizabeth University Hospital - PPDS, Glasgow
  - Raigmore Hospital - PPDS, Inverness
  - The Royal London Hospital, London
  - The National Hospital for Neurology & Neurosurgery, London, GT LON
  - University of Nottingham, Nottingham
  - Peninsula College of Medicine and Dentistry, Plymouth
  - Salford Royal Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing